CLINICAL TRIAL: NCT06979453
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Deucravacitinib in Adolescent Participants (12 Years to Less Than 18 Years) With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Drug Levels of Deucravacitinib (BMS-986165) in Adolescent Participants With Moderate to Severe Plaque Psoriasis
Acronym: POETYK-PsO-Ped
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-1128; 2023-506296-97 (Other: EU CTR); U1111-1289-8030 (Other: WHO)
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Rash; Itch; Teen; Dermatology; Derm; POETYK-PsO-Peds-1
MeSH Terms: conditions — Psoriasis; Exanthema; Pruritus | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Administration of Deucravacitinib (Active Comparator)
  Interventions: Drug: Deucravacitinib
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165
  Arms: Administration of Deucravacitinib
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and drug levels of Deucravacitinib (BMS-986165) in adolescent participants with moderate to severe plaque psoriasis

ELIGIBILITY:
Inclusion Criteria

* Participants must have stable plaque psoriasis for 6 months or more prior to Screening.
* Participants must have moderate to severe psoriasis defined by:.

  i) Psoriasis Area and Severity Index (PASI) ≥ 12, at screening visit and Day 1.

ii) Static Physician's Global Assessment (sPGA) ≥ 3, at screening visit and Day 1.

iii) Body Surface Area (BSA) ≥ 10% involvement, at screening visit and Day 1.

- A female (as assigned at birth) participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:.

i) Is not an individual of childbearing potential (IOCBP).

ii) Is an IOCBP and using a contraceptive method that is highly effective (with a failure rate of < 1% per year) during the study intervention period and for at least 3 days after discontinuation of the study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction for the same period.

Exclusion Criteria

* Participants must not weigh < 30.0 kg at Screening and Day 1.
* Participants must not have non-plaque psoriasis (ie, guttate, inverse, pustular, erythrodermic, or drug-induced psoriasis) or any skin condition other than plaque psoriasis that could interfere with assessments of treatment effect at Screening or Day 1.
* Participants must not have a history of serious bacterial, fungal, or viral infection requiring hospitalization and intravenous (IV) antimicrobial treatment within 60 days prior to Day 1.
* Participants must not have any untreated bacterial infection within 60 days prior to Day 1.
* Participants must not have any ongoing evidence of chronic bacterial infection (eg, chronic pyelonephritis, chronic osteomyelitis, chronic bronchiectasis).
* Participants must not have herpes simplex/zoster, active tuberculosis (TB), hepatitis C virus (HCV), hepatitis B virus (HBV), human immunodeficiency virus (HIV) infection-related exclusions.
* Participants must not have received live vaccines or BCG within 60 days prior to Day 1 or plans to receive a live vaccine during the study, or within 60 days after completing study intervention.
* Participants must not have had any prior exposure to deucravacitinib.
* Participants must not have received any medication that is specifically prohibited.
* Participants must not have a laboratory finding that is exclusionary.
* Participants must not have any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, psychiatric, neurologic, immunologic, or local active infection/infectious illness) that, in the investigator's judgment or after consultation with the Sponsor's Medical Monitor, will substantially increase the risk to the participant if he or she participates in the study.
* Participants must not have cancer or history of cancer (solid organ or hematologic including myelodysplastic syndrome) or lymphoproliferative disease within the previous 5 years.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 366 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2029-10-12 (Estimated); Study Completion 2034-08-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving at least 75% improvement in Psoriasis Area and Severity Index (PASI 75) | At week 16
Number of participants achieving a static Physicians Global Assessment (sPGA) score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline | At week 16

SECONDARY OUTCOMES:
Number of participants achieving at least 90% improvement in PASI (PASI 90) | At week 16
Change from baseline in PASI | At week 16
Change from baseline in body surface area (BSA) involvement | At week 16
Change from baseline in worst itch numeric rating scale (WI-NRS) | At week 16
Number of participants achieving ≥ 4 improvement from baseline in the WI-NRS score (in participants with baseline score ≥ 4) | At week 16
Change from baseline in Children's Dermatology Life Quality Index (CDLQI) score | At week 16
Number of participants achieving CDLQI 0/1 (among participants with a baseline CDLQI score ≥ 2) | At week 16
Number of participants with treatment emergent adverse events | Up to 5 years
Number of participants with serious adverse events | Up to 5 years
Number of participants with clinically significant changes in laboratory parameters | Up to 5 years
Number of participants with clinically significant changes in physical examinations | Up to 5 years
Number of participants with clinically significant changes in vital signs | Up to 5 years
Number of participants with protective titers of antibodies to measles | At week 16
Number of participants with protective titers of antibodies to tetanus | At week 16
Number of participants with protective titers of antibodies to pertussis | At week 16
Body weight | Up to 5 years
Height | Up to 5 years
Sexual maturation | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (114):
- United States (39):
  - Local Institution - 0261, Birmingham, Alabama
  - Local Institution - 0041, Birmingham, Alabama
  - Local Institution - 0053, Phoenix, Arizona
  - Local Institution - 0025, Fountain Valley, California
  - Local Institution - 0090, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - Local Institution - 0077, Sacramento, California
  - Golden State Dermatology - Walnut Creek - Ygnacio Valley Road, Walnut Creek, California
  - Paradigm Clinical Research, LLC, Wheat Ridge, Colorado
  - Local Institution - 0021, Clearwater, Florida
  - Life Clinical Trials, Margate, Florida
  - Skin Research of South Florida, Miami, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Palm Harbor Dermatology PA d/b/a TrueBlue Clinical Research, Tampa, Florida
  - Dermatology Affiliates Research Institute, Atlanta, Georgia
  - Advanced Medical Research, PC., Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Local Institution - 0262, Murray, Kentucky
  - Local Institution - 0202, Metairie, Louisiana
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - Kuchnir Dermatology & Dermatologic Surgery, Milford, Massachusetts
  - Local Institution - 0095, Detroit, Michigan
  - Local Institution - 0233, Columbia, Missouri
  - Local Institution - 0266, Lee's Summit, Missouri
  - Local Institution - 0052, Las Vegas, Nevada
  - Local Institution - 0166, The Bronx, New York
  - Hickory Dermatology Research Center, Hickory, North Carolina
  - Apex Clinical Research Center - Canton, Canton, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Paddington Testing Company, Philadelphia, Pennsylvania
  - ObjectiveHealth - Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - Belle Meade Dermatology Research, Nashville, Tennessee
  - Local Institution - 0268, Austin, Texas
  - Local Institution - 0267, Cedar Park, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Local Institution - 0045, Norfolk, Virginia
  - Frontier Derm Partners, Mill Creek, Washington
  - Local Institution - 0264, Spokane, Washington
- Argentina (6):
  - Local Institution - 0115, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0119, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0149, Buenos Aires
  - Local Institution - 0221, Buenos Aires
  - Local Institution - 0250, Buenos Aires
  - Local Institution - 0154, Buenos Aires
- Belgium (4):
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-Capitale, Région de
  - Local Institution - 0210, Brussels, Bruxelles-Capitale, Région de
  - UZ Gent, Ghent, Oost-Vlaanderen
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Brazil (5):
  - Local Institution - 0137, Salvador, Estado de Bahia
  - Local Institution - 0182, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0136, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0140, Barretos, São Paulo
  - Local Institution - 0163, Ribeirão Preto, São Paulo
- Canada (8):
  - Local Institution - 0241, Edmonton, Alberta
  - Local Institution - 0164, Winnipeg, Manitoba
  - Skincare Studio, St. John's, Newfoundland and Labrador
  - DermEffects, London, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - AvantDerm, Toronto, Ontario
  - Local Institution - 0240, Toronto, Ontario
  - Local Institution - 0142, Montreal, Quebec
- China (9):
  - Beijing Children's hospital, Capital Medical University, Beijing, Beijing Municipality
  - Local Institution - 0222, Beijing, Beijing Municipality
  - Local Institution - 0226, Shenzhen, Guangdong
  - Local Institution - 0255, Handan, Hebei
  - Local Institution - 0227, Zhengzhou, Henan
  - Local Institution - 0265, Jinan, Shandong
  - Local Institution - 0131, Shanghai, Shanghai Municipality
  - Local Institution - 0228, Chengdu, Sichuan
  - Local Institution - 0224, Hangzhou, Zhejiang
- Colombia (4):
  - Local Institution - 0225, Medellín, Antioquia
  - Local Institution - 0124, Medellín, Antioquia
  - Local Institution - 0167, Barranquilla, Atlántico
  - Local Institution - 0125, Bogota, Cundinamarca
- Germany (5):
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - BAG Drs. Med. Quist PartG, Mainz, Rhineland-Palatinate
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
- Hungary (2):
  - Local Institution - 0203, Szeged, Csongrád megye
  - Clinexpert Kft., Budapest, Pest County
- Mexico (8):
  - Local Institution - 0238, Zapopan, Jalisco
  - Local Institution - 0253, Mexico City, Mexico City
  - Local Institution - 0155, Monterrey, Nuevo León
  - Local Institution - 0259, Chihuahua City
  - Local Institution - 0257, Mérida
  - Local Institution - 0237, Puebla City
  - Local Institution - 0258, Toluca
  - Local Institution - 0096, Veracruz
- Poland (7):
  - Local Institution - 0177, Lublin, Lublin Voivodeship
  - FutureMeds - Targowek, Warsaw, Masovian Voivodeship
  - SPECDERM Poznanska sp.j., Bialystok, Podlaskie Voivodeship
  - "DERMED" Centrum Medyczne Sp. z o.o., Lodz
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Klinika Ambroziak Dermatologia, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
- Puerto Rico (3):
  - Local Institution - 0254, Bayamón
  - Local Institution - 0008, Caguas
  - Local Institution - 0012, San Juan
- Romania (6):
  - Local Institution - 0174, Bucharest, București
  - Local Institution - 0249, Bucharest, București
  - Local Institution - 0213, Bucharest, București
  - Policlinica Providența, Iași
  - Centrul de Medicina de Familie, Iași
  - New Derm Clinical SRL, Timișoara
- Spain (4):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [Barcelona]
  - Grupo Pedro Jaén, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
- Taiwan (4):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06979453.html